CLINICAL TRIAL: NCT04207190
Title: Phase 1/1b Trial of Talazoparib and Gemtuzumab Ozogamicin in Adult Patients With Relapsed and/or Refractory Acute Myeloid Leukemia
Brief Title: Talazoparib and Gemtuzumab Ozogamicin for the Treatment of CD33 Positive Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 435819; NCI-2019-07826 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 435819 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-12-10; First posted 2019-12-20 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (talazoparib, gemtuzumab ozogamicin) (Experimental): Patients receive talazoparib PO daily on days 1-21 and gemtuzumab ozogamicin IV over 2 hours on days 1, 4, and 7 or day 1 for patients who CR/CRi after cycles 1 or 2. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemtuzumab Ozogamicin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Talazoparib; Drug: Talazoparib Tosylate

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673
Drug: Talazoparib Tosylate — Given PO
  Other Names: Talzenna

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of talazoparib given together with gemtuzumab ozogamicin and to see how well they work in treating patients with CD33 positive acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory). Talazoparib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Gemtuzumab ozogamicin is a protein (antibody) combined with a chemotherapy drug which specifically targets acute myeloid leukemia cells expressing a marker (CD33). Adding talazoparib to the gemtuzumab ozogamicin therapy may lead to an increased effectiveness in treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of talazoparib given in combination with gemtuzumab ozogamicin therapy in adult patients with relapsed and/or refractory acute myeloid leukemia (AML).

II. Determine the overall response rate (ORR consisting of complete remission [CR] or complete remission with incomplete hematologic recovery [CRi]) of combination therapy with talazoparib and gemtuzumab ozogamicin in patients with relapsed and/or refractory AML.

SECONDARY OBJECTIVE:

I. Evaluate the preliminary anti-leukemic efficacy of talazoparib given in combination with gemtuzumab ozogamicin as determined by complete remission (CR) rate, best response rate (CRi + partial remission [PR]), duration of remission, leukemia-free survival (LFS), transfusion independence (TI), and overall survival (OS) in patients treated with this combination therapy.

EXPLORATORY OBJECTIVES:

I. Evaluate the efficacy of talazoparib given in combination with gemtuzumab ozogamicin on minimal residual disease (MRD) in treated patients.

II. Evaluate mechanistic biomarkers including levels of PARP inhibition and deoxyribonucleic acid (DNA) damage effects in peripheral blood and marrow samples from patients treated with combination therapy.

III. Evaluate quality of life (QOL) of patients with relapsed/refractory AML treated with talazoparib and gemtuzumab ozogamicin.

IV. Evaluate the number of patients able to proceed onto subsequent hematopoietic stem cell transplantation (HSCT) following combination therapy.

OUTLINE: This is a dose-escalation study of talazoparib.

Patients receive talazoparib orally (PO) daily on days 1-21 and gemtuzumab ozogamicin intravenously (IV) over 2 hours on days 1, 4, and 7 or day 1 for patients who CR/CRi after cycles 1 or 2. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status between 0-1
* Creatinine =< 1.5 x upper limit of normal (ULN) or calculated creatinine clearance (Cockcroft and Gault ) > 30 mL/min (performed on plasma unless otherwise indicated)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (performed on plasma unless otherwise indicated)
* Direct bilirubin < 1.5 mg/dL (performed on plasma unless otherwise indicated)
* Left ventricular ejection fraction (LVEF) >= 40% as assessed by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan performed within 28 days of enrollment
* Diagnosis of CD33+ acute myeloid leukemia (AML) with evidence of >= 5% myeloblasts in the bone marrow, peripheral blood, or in an extramedullary site by pathology. Any CD33 receptor expression level > 0.01% by institute flow cytometric analysis will suffice
* Relapsed or refractory disease, defined as:

  * Any bone marrow relapse after allogeneic HSCT: subjects must be at least 1 month from HSCT at the time of screening and off immunosuppressive medication for at least 2 weeks at time of initial treatment (with the exception of low-dose steroids =< 20 mg prednisone equivalent) and have no active graft versus (vs.) host disease (GVHD)
  * AML with no prior CR/CRi after at least 1 prior cycle of remission induction chemotherapy (i.e. cytarabine or hypomethylating based regimen(s) allowed)
  * AML recurring after prior CR/CRi, which was achieved following at least one prior chemotherapy cycle (i.e. cytarabine or hypomethylating based regimen(s) allowed)
* Peripheral white blood cell (WBC) counts <25,000/mcL. Patients are allowed to receive hydroxyurea and/or leukapheresis to control and maintain WBC count prior to enrollment and can continue on hydroxyurea through Cycle 1 Day 28 or until first disease assessment
* Participants of childbearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Acute promyelocytic leukemia (APL, FAB M3) with t(15-17) and/or evidence of promyelocytic leukemia/retinoic acid receptor alpha (PML-RAR alpha)
* Blast phase of prior chronic phase chronic myeloid leukemia with t(9;22)
* Receipt of chemotherapy (except for hydroxyurea), radiotherapy, or investigational drug therapy within 2 weeks prior to treatment on study or those who have not recovered from adverse events due to agents administered > 2 weeks earlier
* Known active central nervous system involvement; patients who have a history of central nervous system (CNS) disease which has been effectively treated as defined by at least one negative cerebrospinal sample prior to screening are eligible
* Active uncontrolled malignancy requiring ongoing chemotherapy and/or radiation. Examples of eligible patients include individuals with a prior history of malignancy treated with curative intent with no current evidence of active disease such as:

  * Subjects with stage I breast cancer that has been completely and successfully treated, requiring no therapy or only anti-hormonal therapy
  * Subjects with T1N0M0 or T2N0M0 colorectal cancer who have been completely and successfully resected and who are disease-free for > 2 years prior to screening
  * Subjects with indolent prostate cancer, defined as clinical stage T1 or T2a, Gleason score =< 6, and prostate specific antigen (PSA) < 10 ng/mL, requiring no therapy or only anti-hormonal therapy
  * Subjects with a history of basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix, fully resected, and with no evidence of active disease
  * Other prior or concurrent malignancies will be considered on a case-by-case basis after discussion with the principal investigator (PI)
* Uncontrolled current medical illness including, but not limited to:

  * Severe cardiac disorder (symptomatic congestive heart failure requiring treatment, chronic unstable angina pectoris, myocardial infarction, cardiac arrhythmia, torsades de pointes,
  * Neurologic impairment (cerebrovascular accident, transient ischemic attack)
  * Severe pulmonary disorder (e.g. DLCO of 65% or less or a forced expiratory volume in 1 second [FEV1]) of 65% of less)
  * Moderate hepatic impairment with total bilirubin >1.5 x upper limit of normal (ULN),
  * Eastern Cooperative Oncology (ECOG ) Performance Status ≥ 2,
  * Any other psychiatric illness/social situations that in the opinion of the investigator would limit compliance with study requirements
* Known malabsorption syndrome or other condition that may impair the absorption of the study drug and/or inability and/or unwillingness to swallow capsules
* Uncontrolled active systemic fungal, bacterial, viral, or other infection with patient still exhibiting ongoing signs and symptoms due to infection despite appropriate anti-infective therapy at time of screening
* Pregnant or breastfeeding female participants
* Known active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening which requires therapy
* Presence of grade II-IV acute or extensive chronic GVHD at time of screening
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug including, but not limited to, medical, psychological, familial, social or geographical considerations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 28 days
  Will identify the maximum tolerated dose of talazoparib in combination with gemtuzumab ozogamicin. The maximum dose level where 1 or fewer dose limiting toxicities (DLTs) are observed in 6 patients will be defined as the recommended phase 2 dose.
Overall response rate (ORR) | Up to 12 months post treatment
  ORR will consist of complete remission (CR), complete remission with incomplete hematologic recovery (CRi) of combination therapy with talazoparib and gemtuzumab ozogamicin. Will be estimated by a 90% confidence interval obtained by Jeffrey's prior method.

SECONDARY OUTCOMES:
Complete remission rate | Up to 12 months post treatment
  The complete remission will be estimated with 90% confidence intervals obtained by Jeffrey's prior method.
Best response rate | Up to 12 months post treatment
  Best response rate will consist of CRi and partial remission (PR).
Duration of remission | Up to 12 months post treatment
  Duration of response will be estimated using standard Kaplan-Meier methods, where estimates of the median will be obtained with 90% confidence intervals.
Leukemia-free survival (LFS) | Up to 12 months post treatment
  LFS will be estimated using standard Kaplan-Meier methods, where estimates of the median will be obtained with 90% confidence intervals.
Transfusion independence rate | Up to 12 months post treatment
  Transfusion independence rate will be estimated with 90% confidence intervals obtained by Jeffrey's prior method.
Hematopoietic stem cell transplantation (HSCT) rates | Up to 12 months post treatment
  HSCT will be estimated with 90% confidence intervals obtained by Jeffrey's prior method.
Overall survival (OS) | Up to 12 months post treatment
  OS will be estimated using standard Kaplan-Meier methods, where estimates of the median will be obtained with 90% confidence intervals.
Incidence of adverse events (AEs) | Up to 30 days post treatment
  The observed AEs, serious AEs (SAEs), DLTs, and toxicities will be summarized by dose level and grade using frequencies and relative frequencies. AEs, SAEs, DLTs, and toxicity rates will be estimated with 90% confidence intervals obtained using Jeffrey's prior method.

CONTACTS AND LOCATIONS:
Overall Officials: Eunice S Wang, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York